CLINICAL TRIAL: NCT05358964
Title: Family Health Histories: Creating a Culturally Tailored Tool to Reduce Health Disparities in the African American Community
Brief Title: Family Health Histories: Creating a Culturally Tailored Tool to Reduce Health Disparities in the Black Community
Acronym: FHH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Michigan State University (Other)
Responsible Party: Principal Investigator, Kent Key, Assistant Professor, Michigan State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 00005570
Record Dates: First submitted 2022-03-14; First posted 2022-05-03 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Hereditary Diseases
MeSH Terms: conditions — Genetic Diseases, Inborn

STUDY DESIGN:
Intervention Model Description: Participants assigned to the AFFHEP will receive a culturally tailored Family Health History Tool designed specifically for African Americans. The Control group will receive the Genetic Alliance Does it Run in the Family Toolkit
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- African American Family Health History Education Program (Experimental): The AAFHHEP arm is an intervention to increase utilization of FHH and increase preventative screening. This tool will be culturally tailored by African Americans for African Americans.
  Interventions: Behavioral: African American Family Health History Education Program
- Genetic Alliance: Does it run in the family (Active Comparator): The Genetic Alliance Does it run in the family is an existing family health history tool kit generalized to all racial groups. This tool is widely available via the internet.
  Interventions: Behavioral: African American Family Health History Education Program

INTERVENTIONS:
Behavioral: African American Family Health History Education Program — The AAFHHEP arm is an intervention to increase utilization of FHH and increase preventative screening. This tool will be culturally tailored by African Americans for African Americans.
  Other Names: AAFHHEP

SUMMARY:
The understanding, utilization and uptake of Family Health History is essential to the prevention of health disparities in the African American community. Creating a culturally tailored Family Health History tool, co-developed by members of the African American community will inform, educate and empower African Americans about health issues related to their family genealogy. Applying the knowledge gained via Family Health Histories to increase preventative behaviors including screenings thus linking people to needed health services to prevent the onset of disease and illness.

DETAILED DESCRIPTION:
African Americans (AA) suffer disproportionately across most health disparities (HD). Preventative behaviors including screenings can inform proactive measures to address many HD which include: diabetes, heart disease, high blood pressure, stroke, HIV, STDs/STIs, cancer, and cardiovascular disease, most of which can be prevented.1-3 Evidence suggests that a lack of general health literacy (HL) and racially appropriate health communication strategies may contribute to the consistent high rates of health disparities in the AA community. Family Health Histories (FHH), which describe genetic and other familial contributions to health, have been identified as an effective tool for prevention and early detection and screenings. The underutilization of FHHs in AA communities negatively impacts screening and preventative measures that could prevent the onset of disease, illness and ultimately death.4 Although many FHH toolkits have been created to assist families in gathering FHH information, these tools typically are mostly focused for the general population and do not account for the cultural and ethnic nuances, communication preference and health literacy levels of the African American community.4 The failure to effectively engage AA in the creation and conception of culturally relevant FHH tools and activities to date likely contributes to their underutilization in this population.

The objective of this K01 is to develop culturally appropriate FHH tools designed for broad understanding and uptake in AA communities. The central hypothesis of this proposal is that, using a community based participatory research (CBPR) approach, co-development of a culturally appropriate FHH toolkit will increase the utility and engagement of AA families in FHH activities; increase effective health communication within the family structure; and increase the health literacy of participants in a multifaceted effort to reduce and ultimately eliminate racial and ethnic health disparities. Flint is an ideal community in which to conduct this participatory research because the recent events of the Flint Water Crisis have created interest in genetics and FHH in the AA community as a result of community concern around the generational impacts of bacteria and lead exposure on health. Therefore, we will have partners within AA communities in Flint who will be motivated to partner with us to develop these tools for Flint and for other minority communities.

This career development award is being submitted by Dr. Kent Key, a candidate with extensive experience in CBPR and a solid foundation in qualitative and health disparities research. To reach his long term goal of becoming an R01-funded researcher in CBPR to reduce health disparities by increasing health literacy and using effective health communication strategies to reduce and ultimately eliminate racial health disparities for African-American populations, this K01 will provide additional training in the following areas: (1) intervention development and design and conduct of randomized trials, (2) health communication models, (3) health literacy promotion, (4) CBPR approaches to Genomics and Genetics, (5) biostatistics, (6) grant-writing.

ELIGIBILITY:
Inclusion Criteria:

* Self Identify as African American; age 18 and older, English speaking

Exclusion Criteria:

* Non English speaking, non African American, younger than 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-03-30 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Use of Family Health History with Family | 3 month
  We will evaluate the length of conversations (minutes per month) with family using a modified Genetic Alliance Assessment
Use of Family Health History with Physician | 3 months
  We will evaluate the length of conversations (minutes per month) with physician using a modified Genetic Alliance Assessment
Quality of Family Health History Discussions | 3 months
  We will evaluate the quality of conversations using the Genetic Alliance Assessment
Quality of Family Health History Discussions | 6 months
  We will evaluate the quality of conversations using the Genetic Alliance Assessment
Acceptability: End of Intervention/Treatment Questionnaire | 3 months
  End of Intervention/Treatment Questionnaire: This is a descriptive measure, positive experiences described meaning higher acceptability
Acceptability: End of Intervention/Treatment Questionnaire | 6 months
  End of Intervention/Treatment Questionnaire: This is a descriptive measure, positive experiences described meaning higher acceptability
Feasibility: End of Intervention/Treatment Questionnaire | 3 months
  End of Intervention/Treatment Questionnaire: This is a descriptive measure, positive experiences described meaning higher acceptability
Feasibility: End of Intervention/Treatment Questionnaire | 6 months
  End of Intervention/Treatment Questionnaire: This is a descriptive measure, positive experiences described meaning higher acceptability
Acceptability: Client Satisfaction Questionnaire (CSQ-8-R) | 3 months
  CSQ-8-R: scores range from 8-32, higher scores indicating higher satisfaction
Acceptability: Client Satisfaction Questionnaire (CSQ-8-R) | 6 months
  CSQ-8-R: scores range from 8-32, higher scores indicating higher satisfaction
Feasibility: Client Satisfaction Questionnaire (CSQ-8-R) | 3 months
  CSQ-8-R: scores range from 8-32, higher scores indicating higher satisfaction
Feasibility: Client Satisfaction Questionnaire (CSQ-8-R) | 6 months
  CSQ-8-R: scores range from 8-32, higher scores indicating higher satisfaction

SECONDARY OUTCOMES:
Satisfaction with Family Health History | 3 months
  We will evaluate satisfaction using the the Client Satisfaction Questionnaire (CSQ-8-R)
Satisfaction with Family Health History | 6 months
  We will evaluate satisfaction using the the Client Satisfaction Questionnaire (CSQ-8-R)
Understandability | 3 months
  We will evaluate understandability using the Health Literacy Questionnaire (HLQ)
Understandability | 6 months
  We will evaluate understandability using the Health Literacy Questionnaire (HLQ)
Number of screenings requested | 3 months
  We will evaluate number of screenings requested using the Family Health Communication Quotient (FHCQ)
Number of screenings requested | 6 months
  We will evaluate number of screenings requested using the Family Health Communication Quotient (FHCQ)

OTHER OUTCOMES:
Health literacy | 3 months
  We will evaluate health literacy using the Health Literacy Questionnaire (HLQ)
Health literacy | 6 months
  We will evaluate health literacy using the Health Literacy Questionnaire (HLQ)
Health communication | 3 months
  We will evaluate health communication using the Health Literacy Questionnaire (HLQ)
Health communication | 6 months
  We will evaluate health communication using the Health Literacy Questionnaire (HLQ)

CONTACTS AND LOCATIONS:
Overall Officials: Kent D Key, PhD, Principal Investigator — Michigan State University
Locations (1):
- Michigan State University, Flint, Michigan, United States

IPD SHARING:
Plan to Share IPD: No
We will not share individual participant data with other researchers. Will will only share data results and summarized data via presentations and manuscript publications.

REFERENCES:
- [Derived] Key KD, Lewis L, Blanchard C, Sikorskii A, Patel M, Lucas T, Henry Akintobi T, Bailey S, Loney EH, Johnson JE. Study protocol: Exploring the use of Family Health Histories in the African American community to reduce health disparities in Flint, Michigan. Res Sq [Preprint]. 2024 Apr 1:rs.3.rs-4131949. doi: 10.21203/rs.3.rs-4131949/v1. PMID 38645135